CLINICAL TRIAL: NCT00566670
Title: Protein Intake, Nutrition and Cardiovascular Disease in Stage 5 Chronic Kidney Disease (CKD)
Brief Title: Protein, Nutrition and Cardiovascular Disease in Stage 5 Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Srinvasan Beddhu, MD, University of Utah
Other Study IDs: IRB_00024816; R01DK077298 (NIH)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 30 ml of blood drawn four times (months 1, 6, 12 and 18) for plasma/serum/DNA samples.
  Urine Collection: If patients are making more than ½ cup (200 ml) of urine a day.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation (all participants): Stage 5 Chronic Kidney Disease and hemodialysis patients

SUMMARY:
National Kidney Foundation guidelines recommend a dietary protein intake of 1.2 grams per kilogram per day (g/kg/d) in hemodialysis patients. However, it is unclear whether consumption of high amounts of protein in dialysis patients has beneficial or harmful nutritional and cardiovascular effects in this population. High protein intake might improve nutritional status, but it has been argued that the state of low muscle mass, small body size and low serum protein levels is not the result of decreased dietary intake, rather a result of hypercatabolism induced by metabolic acidosis, inflammation and oxidative stress.

The specific aims of this study are to examine in a prospective cohort of hemodialysis patients the longitudinal associations of absolute total protein intake or dietary protein intake with muscle mass and arterial stiffness.

DETAILED DESCRIPTION:
It is hypothesized that in the dialysis population overall: (1) Protein intake is a major determinant of muscle mass while inflammation, oxidative stress and metabolic acidosis play a lesser role; (2) Malnutrition is not an uremic cardiovascular risk factor hence low protein intake does not cause cardiovascular disease; and (3) In the other extreme, high protein intake is also not a major cause of cardiovascular disease since high serum phosphorus associated with high protein intake can usually be controlled by the use of phosphorus binders in routine clinical practice.

The specific aims of this proposal are to examine in a prospective cohort of hemodialysis patients the longitudinal associations of absolute total protein intake (TPI) in grams/day, or dietary protein intake (DPI) normalized to body weight in grams/kilogram/day) with

1. Nutritional status (mid-thigh muscle mass as measured by Magnetic Resonance Imaging ) and functional status (6-min walk) and
2. Arterial stiffness (aortic pulse wave velocity)

Understanding the relationship between protein intake with body composition (muscle mass) and intermediate cardiovascular outcomes (arterial stiffness) in stage 5 CKD patients in hemodialysis is of great scientific and practical significance

ELIGIBILITY:
Inclusion Criteria:

* Adult stage 5 chronic kidney disease patients, on dialysis for at least 3 months.
* Urine output > 200 mL/day

Exclusion Criteria:

* Patients with persistent volume overload (substantial pedal edema) despite attempts at achieving dry weight
* Patients with inability to walk or who use a wheel-chair with reduced mid-thigh muscle mass
* Persons with pacemakers, cochlear implants, or other prohibitive conditions for magnetic resonance imaging
* Atrial fibrillation
* Patients who are unlikely or unable (in the opinion of the nephrologists, nurses or dieticians taking care of the patient) to comply with research protocol
* Patients with symptomatic heart failure, current active malignancy (excluding squamous and basal cell skin cancers), active AIDS, chronic lung disease requiring supplemental oxygen therapy and cirrhosis
* Patients enrolled in interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of Utah Dialysis Program patients, and Vanderbilt University dialysis patients.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2007-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Correlation of muscle mass with protein intake | Baseline and 18 months
  Mid-thigh muscle mass measured by magnetic resonance imaging

SECONDARY OUTCOMES:
Correlation of arterial stiffness with protein intake | Baseline and 18 months
  Radial artery stiffness measured by pulse wave velocity and pulse wave assessment

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Beddhu, M.D, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Vanderbilt University Medical Centet, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah